CLINICAL TRIAL: NCT05157490
Title: Preoperative Mindfulness Training for Minimally Invasive Hysterectomy
Brief Title: Preoperative Mindfulness: Minimally Invasive Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Howard University (Other); Headspace Meditation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-12609
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training (Experimental): Completion of guided meditations in the preoperative time period, at least 3 sessions per week, leading up to surgery
  Interventions: Behavioral: Mindfulness training
- Control (No Intervention): Standard pre- and postoperative medications will be given to the patients.

INTERVENTIONS:
Behavioral: Mindfulness training — Guided meditations in the preoperative time period, at least 3 sessions per week, leading up to surgery
  Arms: Mindfulness training

SUMMARY:
This is a randomized control trial investigating the effects of a preoperative mindfulness intervention on postoperative pain, quality of recovery and stress scores in women undergoing minimally invasive hysterectomy. The mindfulness intervention will be delivered via the application Headspace™. The study team hypothesizes that mindfulness practiced in the form of meditation delivered via an internet application will lead to reduced pain scores on postoperative day 1.

DETAILED DESCRIPTION:
Pain is a subjective experience influenced by both physical and psychosocial factors.

Postoperative pain can be difficult to treat, frequently leading to underassessment, undertreatment, decreased patient satisfaction and decreased quality of life. Historically efforts have focused on pharmacologic treatments, with opioids commonly being used to manage acute postoperative pain. Overprescribing of opioids remains prevalent despite now well studied adverse outcomes including increased risk for longer length of inpatient stay, future hospitalizations, and risk of dependence. Particularly in the setting of the opioid epidemic, non-pharmacologic interventions for pain management have become more attractive to practitioners and patients alike.

Psychosocial aspects of pain including catastrophizing, fear, and negative emotions can be targeted by interventions such as mindfulness training, hypnotic suggestion, and psychoeducation. Mindfulness meditations have been shown to engage mechanisms distinct from placebo by attenuating the subjective experience of pain and may be particularly effective when used in combination with pharmacologic analgesia. Mindfulness based interventions have been better studied in the setting of chronic pain with limited data available in the setting of acute pain. In the gynecology literature, dispositional mindfulness was demonstrated to have a positive effect on postoperative pain scores, but no studies to date have examined the effect of pre-procedure mindfulness interventions specifically on postoperative pain. In addition, those studies which exist have focused on populations that are majority non-Hispanic white and have utilized sessions conducted with trained social workers. The investigator team believes there is a unique opportunity to investigate the effects of mindfulness interventions delivered via a systematically reviewed internet application in an urban academic tertiary care center on postoperative pain. This is the first study to examine the effect of preoperative mindfulness training on the recovery process, pain and stress associated with hysterectomy and could represent a low cost, low risk intervention in order to improve perioperative well-being.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo minimally invasive hysterectomy
* Fluency in English and/or Spanish
* Access to a device capable of running the Headspace application (smart phone or computer)

Exclusion Criteria:

* Minors
* Hearing impairment
* Inability to access Headspace app
* Inability to complete baseline or postoperative surveys: Perceived Stress Scale-10 (PSS-10) or Quality of Recovery-15 (QOR-15) surveys

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Pain score | 1 day postoperatively
  Pain scores will be measured on postoperative Day 1 (POD1) using the validated Numeric Pain Rating Scale. The Numeric Pain Rating scale is an 11-point pain intensity rating scale (PI-NRS) ranging from 1-10, where 0 = "No pain" and 10 = "Worst possible pain" such that higher scores are associated with greater pain severity/intensity. Scores will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
Pain score | 7 days postoperatively
  Pain scores will also be measured on postoperative Day 7 (POD7) using the validated Numeric Pain Rating Scale. The Numeric Pain Rating scale is an 11-point pain intensity rating scale (PI-NRS) ranging from 1-10, where 0 = "No pain" and 10 = "Worst possible pain" such that higher scores are associated with greater pain severity/intensity. Scores will be summarized by study arm using basic descriptive statistics.
Quality of Recovery | 1 day and 7 days postoperatively (POD1 and POD7)
  Quality of Recovery will be assessed on POD1 and POD7 using the Quality of Recovery-15 (QoR-15) scale. The QoR-15 is a patient-reported tool measuring post-surgical recovery, using 15 questions across domains such as pain, physical comfort, emotional state, physical independence, and psychological support over the prior 24-hour period. Each question on the QoR-15 is rated using an 11-point numerical rating scale ranging from 0 = "None of the time" to 15 = "All of the time" yielding an overall possible scoring range of 0-150. The final five items are reverse coded. Higher scores are associated with better quality of recovery. Scores will be summarized by study arm using basic descriptive statistics.
Perceived Stress | 1 day and 7 days postoperatively (POD1 and POD7)
  Perceived stress will be assessed on POD1 and POD7 using the 10-item Perceived Stress Scoring (PSS-10) scale. The PSS-10 presents patients with 10 questions and asks them to rate how often they felt a certain way regarding specific feelings and thoughts over the prior month. Responses are rated using a 4-point Likert scale wherein 0 = "Never," 1 = "Almost never," 2 = "Sometimes," 3 = "Often," and 4 = "Very often" yielding a total overall score of 0-40. Four of the questions/items are reverse coded and their scores are reversed (i.e., 0=4, 1=3, 2=2, 3=1, 4=0). Higher scores are associated with increased feelings of perceived stress and helplessness. Scores will be summarized by study arm using basic descriptive statistics.
Opioid consumption | 1 day and 7 days postoperatively (POD1 and POD7)
  The number of opioid/analgesic tablets used postoperatively will be determined by telephone surveys administered on POD1 and POD7. Results will be summarized by study arm.
Non-analgesic opioid consumption | 1 day and 7 days postoperatively (POD1 and POD7)
  The number of non-analgesic opioid tablets used postoperatively will be determined by telephone surveys administered on POD1 and POD7. Results will be summarized by study arm.
Effect of Meditation Session | Up to 7 days postoperatively
  The effect of meditation sessions will be assessed by dose response based on the number of meditation sessions OR the number of minutes of meditation performed, on pain and quality of recovery scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kari M Plewniak, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center-Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Lin RJ, Reid MC, Liu LL, Chused AE, Evans AT. The Barriers to High-Quality Inpatient Pain Management: A Qualitative Study. Am J Hosp Palliat Care. 2015 Sep;32(6):594-9. doi: 10.1177/1049909114530491. Epub 2014 Apr 11. PMID 24728202
- [Background] Burden M, Keniston A, Wallace MA, Busse JW, Casademont J, Chadaga SR, Chandrasekaran S, Cicardi M, Cunningham JM, Filella D, Hoody D, Hilden D, Hsieh MJ, Lee YS, Melley DD, Munoa A, Perego F, Shu CC, Sohn CH, Spence J, Thurman L, Towns CR, You J, Zocchi L, Albert RK. Opioid Utilization and Perception of Pain Control in Hospitalized Patients: A Cross-Sectional Study of 11 Sites in 8 Countries. J Hosp Med. 2019 Dec 1;14(12):737-745. doi: 10.12788/jhm.3256. Epub 2019 Jul 24. PMID 31339840
- [Background] Liang Y, Turner BJ. National cohort study of opioid analgesic dose and risk of future hospitalization. J Hosp Med. 2015 Jul;10(7):425-31. doi: 10.1002/jhm.2350. Epub 2015 Mar 16. PMID 25772626
- [Background] Houry D, Baldwin G. Announcing the CDC guideline for prescribing opioids for chronic pain. J Safety Res. 2016 Jun;57:83-4. doi: 10.1016/j.jsr.2016.03.007. Epub 2016 Apr 16. PMID 27178083
- [Background] Apkarian AV, Bushnell MC, Treede RD, Zubieta JK. Human brain mechanisms of pain perception and regulation in health and disease. Eur J Pain. 2005 Aug;9(4):463-84. doi: 10.1016/j.ejpain.2004.11.001. Epub 2005 Jan 21. PMID 15979027
- [Background] Wiech K, Tracey I. The influence of negative emotions on pain: behavioral effects and neural mechanisms. Neuroimage. 2009 Sep;47(3):987-94. doi: 10.1016/j.neuroimage.2009.05.059. Epub 2009 May 28. PMID 19481610
- [Background] Zeidan F, Vago DR. Mindfulness meditation-based pain relief: a mechanistic account. Ann N Y Acad Sci. 2016 Jun;1373(1):114-27. doi: 10.1111/nyas.13153. PMID 27398643
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Garland EL, Baker AK, Larsen P, Riquino MR, Priddy SE, Thomas E, Hanley AW, Galbraith P, Wanner N, Nakamura Y. Randomized Controlled Trial of Brief Mindfulness Training and Hypnotic Suggestion for Acute Pain Relief in the Hospital Setting. J Gen Intern Med. 2017 Oct;32(10):1106-1113. doi: 10.1007/s11606-017-4116-9. Epub 2017 Jul 12. PMID 28702870
- [Background] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Background] McClintock AS, McCarrick SM, Garland EL, Zeidan F, Zgierska AE. Brief Mindfulness-Based Interventions for Acute and Chronic Pain: A Systematic Review. J Altern Complement Med. 2019 Mar;25(3):265-278. doi: 10.1089/acm.2018.0351. Epub 2018 Dec 5. PMID 30523705
- [Background] Weston E, Raker C, Huang D, Parker A, Robison K, Mathews C. The Association Between Mindfulness and Postoperative Pain: A Prospective Cohort Study of Gynecologic Oncology Patients Undergoing Minimally Invasive Hysterectomy. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1119-1126.e2. doi: 10.1016/j.jmig.2019.08.021. Epub 2019 Aug 23. PMID 31449907
- [Background] Mani M, Kavanagh DJ, Hides L, Stoyanov SR. Review and Evaluation of Mindfulness-Based iPhone Apps. JMIR Mhealth Uhealth. 2015 Aug 19;3(3):e82. doi: 10.2196/mhealth.4328. PMID 26290327
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Choi JB, Kang K, Song MK, Seok S, Kim YH, Kim JE. Pain Characteristics after Total Laparoscopic Hysterectomy. Int J Med Sci. 2016 Jul 5;13(8):562-8. doi: 10.7150/ijms.15875. eCollection 2016. PMID 27499688
- [Background] Wright JD, Herzog TJ, Tsui J, Ananth CV, Lewin SN, Lu YS, Neugut AI, Hershman DL. Nationwide trends in the performance of inpatient hysterectomy in the United States. Obstet Gynecol. 2013 Aug;122(2 Pt 1):233-241. doi: 10.1097/AOG.0b013e318299a6cf. PMID 23969789
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Baik SH, Fox RS, Mills SD, Roesch SC, Sadler GR, Klonoff EA, Malcarne VL. Reliability and validity of the Perceived Stress Scale-10 in Hispanic Americans with English or Spanish language preference. J Health Psychol. 2019 Apr;24(5):628-639. doi: 10.1177/1359105316684938. Epub 2017 Jan 5. PMID 28810432
- See also: Journal of Applied Social Psychology, 42, 1320-1334. This article provides Normative Data for the PSS-10 from large 2006 and 2009 probability samples of the U.S. — https://www.cmu.edu/dietrich/psychology/stress-immunity-disease-lab/scales/pdf/whos_stressed_jasp_2012.pdf